CLINICAL TRIAL: NCT07045272
Title: Study on the Construction and Effectiveness of a Digital Behavioral Intervention Program for Overweight and Obese Patients Prior to Assisted Reproductive Technology(ART)Treatment
Brief Title: Effectiveness of a Digital Behavioral Intervention Program for Overweight and Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Wang Danni, Associate Professor, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WDanni
Record Dates: First submitted 2025-06-09; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital behavioral intervention (Experimental): A comprehensive intervention program that combines digital technologies，Including interventions for diet, exercise, mood, sleep, etc.
  Interventions: Behavioral: Experimental
- Regular Education Group (No Intervention): Physicians provided only their standard verbal counseling during clinic visits, without any additional interventions.

INTERVENTIONS:
Behavioral: Experimental — The intervention team provides lifestyle guidance to the subjects according to the behavioural intervention programme, and the subjects record information on diet, exercise and weight on the platform on a daily basis. Subjects are required to learn relevant health education knowledge on the platform by themselves, and they can also exchange experience in the group and receive motivational counselling from the instructors.
  Arms: digital behavioral intervention

SUMMARY:
This study applied digital technology to a comprehensive lifestyle intervention strategy to design a digital behavioural intervention programme suitable for weight reduction in overweight obese infertile patients in China, and assessed its intervention effect through a randomised controlled trial.The main questions it aims to answer are:

1) Design and implement a digital behavioural weight loss intervention programme; 2) Evaluate the impact of digital behavioural interventions on weight loss outcomes and health outcomes.

Participants will be randomly assigned to a control group and an intervention group.

The control group will receive only routine health education and the intervention group will receive an 8-week digital behavioural intervention. At the end of the intervention, the follow-up period will be one year for reproductive outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilling the World Health Organization diagnostic criteria for infertility, defined as failure to achieve or sustain a clinical pregnancy after ≥1 year of regular unprotected sexual intercourse among couples of reproductive age;
2. patients aged 20-40 years seeking assisted reproductive technology (ART) treatment;
3. Body mass index (BMI) >=24 kg/m²;
4. Willingness to undergo randomization;
5. Absence of significant comorbidities (e.g., uncontrolled hypertension, diabetes mellitus, malignancies);
6. Commitment to participate in and complete the intervention protocol.

Exclusion Criteria:

1. History of major systemic diseases (e.g., cardiovascular disorders, chronic respiratory diseases) or psychiatric disorders (e.g., schizophrenia, major depressive disorder);
2. Current or prior participation in other clinical trials within the past 3 months;
3. Medical contraindications to physical exercise (e.g., severe osteoarthritis, uncontrolled arrhythmias);
4. Previous weight-loss interventions, including pharmacological therapy (e.g., orlistat, liraglutide) or bariatric surgery.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Weight change | From enrollment to the end of treatment at 8 weeks
Number of oocytes retrieved | up to 16weeks
Number of embryos available for transfer | up to 17 weeks

SECONDARY OUTCOMES:
Percentage of weight loss | From enrollment to the end of treatment at 8 weeks
Body fat content and distribution | From enrollment to the end of treatment at 8 weeks
  using the InBody instrument, which relies on the principle of bioelectrical impedance analysis (BIA) to rapidly assess body composition without radiation exposure.
live birth rate | 2 years
Pregnancy rate | up to 1 year

IPD SHARING:
Plan to Share IPD: Yes